CLINICAL TRIAL: NCT02009930
Title: Assessment of Coronary Artery Calcium in Active Duty Enlisted Military Members With 10 or More Years of Service
Status: Terminated | Type: Observational
Why Stopped: Failure to recruit enough subjects
Sponsor: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Elijah Burton, Radiology Resident, David Grant U.S. Air Force Medical Center
Other Study IDs: FDG20130024H
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Results first posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Atherosclerosis; Plaque, Atherosclerotic
Keywords: Military Active Duty Enlisted; Atherosclerosis; Coronary Artery Calcium (CAC); Cardiovascular; CAC Score; Framingham Score; CT Scan
MeSH Terms: conditions — Atherosclerosis; Plaque, Atherosclerotic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypothesis: Enlisted military members with 10 or more years of service and at least one cardiovascular risk factor will demonstrate a higher risk of future cardiac events as assessed by coronary artery calcium (CAC) scoring than the risk calculated by the Framingham Risk Score.

DETAILED DESCRIPTION:
While the military is making strides towards improving the health and habits of service members, there are many aspects of the military culture that negatively affect the cardiovascular health of military members. Smoking/tobacco use, poor eating habits with Meals Ready-to-eat (MRE) and ready access to fast food establishments on base, inconsistent exercise, the socioeconomic status of enlisted members and the stress of deployment are all factors that contribute to increased risk of cardiovascular disease during military service. Currently the calculation of a patient's Framingham risk score is the most commonly used method of calculating a patient's cardiovascular risk, and this calculation is based on age, smoking history, blood pressure, and lab values and compares it to a general population's risk. By the use of a cardiac computerized topography (CT) scan, a Coronary Artery Calcium (CAC) score can be calculated and used to estimate the degree of atherosclerosis already present in each patient's coronary arteries, and thus establishing their risk of future cardiovascular events. CAC scoring is a more patient-specific way of identifying cardiovascular risk. The purpose of this study is to assess the prevalence of atherosclerosis in enlisted military members with at least 10 years of service and one or more cardiovascular risk factor and to determine if their risk of a cardiovascular event is higher than predicted by the Framingham score. If CAC scoring is demonstrated to be more accurate, particularly if it is more likely to detect risk, it may be used in the future to better risk stratify this population of the military. The CAC results in patients could also be a motivating factor to create changes in the military culture to attempt to mitigate these risks and create a healthier fighting force.

ELIGIBILITY:
INCLUSION Criteria:

Active Duty Military Members with at least 10 years of service

Enlisted Rank

Males 35 years and older OR Females 45 years and older (please note the age difference is due to the fact that female plaque formation with calcification has been shown to lag that of males by about 10 years)

One or More of the Following Risk Factors:

Smoker - at least 5 pack years in the past 5 years (pack year = number of packs per day number of years of smoking)

Diabetic (Fasting glucose of >125 mg/dL on two or more blood draws, or Random Blood Glucose of >200 mg/dL on a single blood draw, or Hemoglobin A1C >6.5%, or previous diagnosis of diabetes listed in the subject's medical record) or Pre-diabetic (Fasting glucose >100 on two or more blood draws or Hgb A1C 5.7-6.4)

Hypertension (Systolic BP > 140 or Diastolic BP >90 or on blood pressure medications or diagnosis of hypertension in medical record)

Waist Circumference > 40 inches for males or >35 inches for females

Hyperlipidemia (LDL>130, HDL<40 for males, HDL <50 for females, Triglycerides >200, on lipid lowering medications and/or diagnosis of hyperlipidemia in medical record)

EXCLUSION Criteria:

Males <35 years old

Women <45 years old (please note the age difference is due to the fact that female plaque formation with calcification has been shown to lag that of males by about 10 years)

Officer Rank - officers are excluded as we are looking at the enlisted culture in the military.

History of any of the following:

Coronary Artery Disease (CAD)

Coronary Artery Bypass Grafting (CABG)

Myocardial Infarction (MI)

Percutaneous Intervention/Stent Placement (PCI)

Angina

Radiotherapy (external beam, brachytherapy, radiopharmaceutical)

Under the care of any of the following types of providers in the past 12 months (As these subjects are at greater risk of having had significant radiation exposure to the chest over the past 12 months):

Radiation/Medical Oncologist

Interventional Radiologist

Cardiologist

Cardiothoracic Surgeon

Vascular Surgeon

Females who think they may be pregnant

Pregnant females

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Active duty military enlisted members with 10 or more years of service
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2013-11-05 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elijah Burton, MD, Principal Investigator — David Grant USAF Medical Center
Locations (1):
- David Grant USAF Medical Center, Travis Air Force Base, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 withdrawn
Groups:
- Coronary Artery Calcium (CAC) / Framingham Risk Score (FRS): Coronary Artery Calcium (CAC) scores are reported as a numerical value and a percentage for age that is then regarded in terms of risk categories. The Framingham Risk Score (FRS) is a standard of care for estimating risk of a cardiovascular event over the next 10 years
Period: Overall Study
Arm/Group | Coronary Artery Calcium (CAC) / Framingham Risk Score (FRS)
Started | 112 (5 withdrawn)
Completed | 107
Not Completed | 5
Not completed — withdrawn | 5

BASELINE CHARACTERISTICS:
Population: 5 withdrawn
Arm/Group | Coronary Artery Calcium (CAC) / Framingham Risk Score (FRS)
Number analyzed (Participants) | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.78505 (5.037647)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 5 withdrawn
  Participants
    Female | 3
    Male | 104
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
More than one cardiovascular risk factor [Count of Participants; unit: Participants] — Population: 5 withdrawn
  Participants | 107

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Atherosclerosis
Description: Percent of active duty enlisted military members with 10 or more years of military service determined to have a prevalence of atherosclerosis based on CAC risk category. The CAC risk category (scale), is derived from the CAC score (i.e., an estimate of the degree of atherosclerosis present in each participant's coronary arteries, reported as a number), and percentage by age to establish risk of future CV events. There are 5 risk categories: Low risk = CAC of 0 and no cardiovascular (CV) risk factors, Low - Moderate risk = CAC of 0 with CV risk factors, Moderate - High risk: CAC 1-100 and percentile for age <75%, High risk = CAC 100-399 or percentile for age >75%, Very high risk = CAC >100 and percentile for age >90% or CAC >400". Low risk is the best outcome, and very high risk is the worst.
Time Frame: within 10 days of CT scan
Measure: Count of Participants; unit: Participants
Groups:
- Coronary Artery Calcium (CAC): Compare CAC risk categories (low, low-mod, mod-high and very high) between groups
Arm/Group | Coronary Artery Calcium (CAC)
Number analyzed (Participants) | 107
Participants | 16
Statistical Analysis 1: Comparison: Coronary Artery Calcium (CAC); Test type: Other; Wilson Method used = 16, 95% CI 2-sided [9.4 to 22.9]

2. Primary Outcome: Rate of Reclassification
Description: Percent/Number of subject that were reclassified from FRS to CAC risk category using CAC scores. The CAC risk category (scale) = CAC score (estimated degree of calcium in coronary arteries, a number) + percentage by age to establish risks of future CV events. There are 5 risk categories: low, low - moderate, moderate - high, very high. The Framingham risk category (scale) = FRS to estimate the risk of a CV event over the next 10 years. The FRS uses age, systolic blood pressure, high-density lipoprotein (HDL) cholesterol level, total cholesterol level, and smoking status to create a score that is converted into a 10-year CV disease risk % that correlates into a risk category: low, moderate, moderate - high risk, very high. For both scales, low is the best and very high is the worst outcome
Time Frame: within 10 days of CT scan
Measure: Count of Participants; unit: Participants
Groups:
- Coronary Artery Calcification (CAC): Compare CAC risk categories (low, low-mod, mod-high and very high) between groups
Arm/Group | Coronary Artery Calcification (CAC)
Number analyzed (Participants) | 107
Participants
  higher risk category | 99
  lower risk category | 5
  same risk category | 3
Statistical Analysis 1: Comparison: Coronary Artery Calcification (CAC); Test type: Other; Only descriptive statistics were calculated (frequency, percent). Inferential statistics were not necessary, nor appropriate

3. Primary Outcome: Compare FRS to the CAC - At Least One Additional Risk Factor
Description: Compare FRS risk category to CAC risk category for enlisted subjects with at least 10 years of service and at least one additional CV risk factor to determine how well the results correlate with one another using the Spearman's Rank Correlation Coefficient. The CAC risk category (scale) = CAC score (estimated degree of calcium in coronary arteries, a number) + percentage by age to establish risks of future CV events. There are 5 risk categories: low, low - moderate, moderate - high, very high. The Framingham risk category (scale) = FRS to estimate the risk of a CV event over the next 10 years. The FRS uses age, systolic blood pressure, high-density lipoprotein (HDL) cholesterol level, total cholesterol level, and smoking status to create a score that is converted into a 10-year CV disease risk % that correlates into a risk category: low, moderate, moderate - high risk, very high. For both scales, low is the best and very high is the worst outcome
Time Frame: within 10 days of CT scan
Population: The data is separated into two rows for each arm. Each row corresponds to a group. Participants were placed into one of the two groups based on certain criteria. Each group has a different number of participants analyzed. The total for both groups (rows) is equal to the overall number of participants analyzed
Measure: Count of Participants; unit: Participants
Groups:
- FRS Risk Category: Compare FRS risk categories (low, moderate, moderate -high, high, and very high) between groups
- CAC Risk Category: Compare CAC risk categories (low, low - moderate, moderate -high, high, and very high) between groups
Arm/Group | FRS Risk Category | CAC Risk Category
Number analyzed (Participants) | 107 | 107
Participants
  at least 1 additional risk factor | 56 | 56
  no additional risk factors | 51 | 51
Statistical Analysis 1: Comparison: FRS Risk Category vs CAC Risk Category; Compare risk categories (FRS and CAC); Test type: Other; p = 0.79, Spearman's Rank Correlation Coefficient — Correlation between FRS and CAC risk categories in participants with at least 1 additional risk factor expressed as a p-value; Correlation between FRS and CAC risk categories in participants with at least 1 additional risk factor. Spearman's rho = 0.04

4. Secondary Outcome: Metabolic Syndrome - Compare FRS to CAC
Description: Compare FRS category and CAC risk category for those meeting and not meeting criteria for metabolic syndrome. Calculate Fisher's Exact test statistic and associated p values to look at the relationship between the presence/absence of metabolic syndrome and the FRS and CAC risk category. The CAC risk category (scale) = CAC score (estimated degree of calcium in coronary arteries, a number) + percentage by age to establish risks of future CV events. There are 5 risk categories: low, low - moderate, moderate - high, very high. The Framingham risk category (scale) = FRS to estimate the risk of a CV event over the next 10 years. The FRS uses age, systolic blood pressure, high-density lipoprotein (HDL) cholesterol level, total cholesterol level, and smoking status to create a score that is converted into a 10-year CV disease risk % that correlates into a risk category: low, moderate, moderate - high risk, very high. For both scales, low is the best and very high is the worst outcome
Time Frame: within 10 days of CT scan
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | FRS Risk Category | CAC Risk Category
Number analyzed (Participants) | 107 | 107
Participants
  metabolic syndrome: number analyzed (Participants) | 23 | 23
  metabolic syndrome: low risk | 19 | 0
  metabolic syndrome: low - moderate / moderate risk | 1 | 18
  metabolic syndrome: moderate - high risk | 3 | 4
  metabolic syndrome: high risk | 0 | 1
  metabolic syndrome: very high risk | 0 | 0
  no metabolic syndrome: number analyzed (Participants) | 84 | 84
  no metabolic syndrome: low risk | 80 | 0
  no metabolic syndrome: low - moderate / moderate risk | 0 | 73
  no metabolic syndrome: moderate - high risk | 4 | 4
  no metabolic syndrome: high risk | 0 | 5
  no metabolic syndrome: very high risk | 0 | 2
Statistical Analysis 1: Comparison: FRS Risk Category; FRS risk category (low, mod, mod-high, high, very high risk); Test type: Other; p = 0.063, Fisher Exact — Relationship between FRS and metabolic syndrome. FRS risk category (low, mod, mod-high, high, very high risk) and metabolic syndrome (presence/absence of metabolic syndrome); Relationship between 2 variables (FRS - each risk category, metabolic syndrome - presence/absence) expressed as a p-value
Statistical Analysis 2: Comparison: CAC Risk Category; CAC risk category (low, low-mod, mod-high, high, very high); Test type: Other; p = 0.21, Fisher Exact — Relationship between CAC and metabolic syndrome. CAC risk category (low, low-mod, mod-high, high, very high risk) and metabolic syndrome (presence/absence of metabolic syndrome); Relationship between 2 variables (CAC - each risk category, metabolic syndrome - presence/absence) expressed as a p-value

5. Secondary Outcome: Living in the Dorms - Compare FRS to CAC
Description: Compare FRS category to CAC risk category for those who lived in the dorms > 5 years and < 5 years. Calculate Fisher's Exact test statistic and associated p values to look at the relationship between those who lived in the dorms > 5 years and < 5 years and the FRS and CAC risk category. The CAC risk category (scale) = CAC score (estimated degree of calcium in coronary arteries, a number) + percentage by age to establish risks of future CV events. There are 5 risk categories: low, low - moderate, moderate - high, very high. The Framingham risk category (scale) = FRS to estimate the risk of a CV event over the next 10 years. The FRS uses age, systolic blood pressure, high-density lipoprotein (HDL) cholesterol level, total cholesterol level, and smoking status to create a score that is converted into a 10-year CV disease risk % that correlates into a risk category: low, moderate, moderate - high risk, very high. For both scales, low is the best and very high is the worst outcome
Time Frame: within 10 days of CT scan
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | FRS Risk Category | CAC Risk Category
Number analyzed (Participants) | 107 | 107
Participants
  > 5 years living in dorms: number analyzed (Participants) | 10 | 10
  > 5 years living in dorms: low risk | 9 | 0
  > 5 years living in dorms: low - moderate / moderate risk | 0 | 7
  > 5 years living in dorms: moderate - high risk | 1 | 1
  > 5 years living in dorms: high risk | 0 | 2
  > 5 years living in dorms: very high risk | 0 | 0
  < 5 years living in dorms: number analyzed (Participants) | 97 | 97
  < 5 years living in dorms: low risk | 90 | 0
  < 5 years living in dorms: low - moderate / moderate risk | 1 | 84
  < 5 years living in dorms: moderate - high risk | 6 | 7
  < 5 years living in dorms: high risk | 0 | 4
  < 5 years living in dorms: very high risk | 0 | 2
Statistical Analysis 1: Comparison: FRS Risk Category; FRS risk categories (low, moderate, mod -high, high, and very high); Test type: Other; p = 0.56, Fisher Exact — Relationship between FRS and living in the dorms. FRS risk category (low, mod, mod-high, high, very high risk) and living in the dorms (< 5 years, > 5 years); Relationship between 2 variables (FRS - each risk category, living in the dorms - <5 years/> 5 years) expressed as a p-value
Statistical Analysis 2: Comparison: CAC Risk Category; CAC risk category (low, low-mod, moderate - high, high, and very high); Test type: Other; p = 0.13, Fisher Exact — Relationship between CAC and living in the dorms. CAC risk category (low, low-mod, mod-high, high, very high risk) and living in the dorms (< 5 years, > 5 years); Relationship between 2 variables (CAC - each risk category, living in the dorms - <5 years/> 5 years) expressed as a p-value

6. Secondary Outcome: Physical Fitness (PT) Failures - Compare FRS to CAC
Description: Compare FRS category to CAC risk category for those with and without PT failures. Calculate Fischer's Exact test statistic and associated p values to look at the relationship between those with and without PT failures and the FRS and CAC risk category. The CAC risk category (scale) = CAC score (estimated degree of calcium in coronary arteries, a number) + percentage by age to establish risks of future CV events. There are 5 risk categories: low, low - moderate, moderate - high, very high. The Framingham risk category (scale) = FRS to estimate the risk of a CV event over the next 10 years. The FRS uses age, systolic blood pressure, high-density lipoprotein (HDL) cholesterol level, total cholesterol level, and smoking status to create a score that is converted into a 10-year CV disease risk % that correlates into a risk category: low, moderate, moderate - high risk, very high. For both scales, low is the best and very high is the worst outcome
Time Frame: within 10 days of CT scan
Population: 1 subject had no data. Data are separated into 2 rows (groups). Participants were placed into 1 of 2 groups based on certain criteria. Each group has a different number of participants. The total for both groups (rows) is equal to the overall number of participants analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | FRS Risk Category | CAC Risk Category
Number analyzed (Participants) | 106 | 106
Participants
  with PT failure: number analyzed (Participants) | 53 | 53
  with PT failure: low risk | 48 | 0
  with PT failure: low - moderate / moderate risk | 0 | 46
  with PT failure: moderate - high risk | 5 | 3
  with PT failure: high risk | 0 | 2
  with PT failure: very high risk | 0 | 2
  without PT failure: number analyzed (Participants) | 53 | 53
  without PT failure: low risk | 50 | 0
  without PT failure: low - moderate / moderate risk | 1 | 44
  without PT failure: moderate - high risk | 2 | 5
  without PT failure: high risk | 0 | 4
  without PT failure: very high risk | 0 | 0
Statistical Analysis 1: Comparison: FRS Risk Category; FRS risk categories (low, moderate, moderate-high, high, and very high); Test type: Other; p = 0.44, Fisher Exact — Relationship between FRS and PT failures. FRS risk category (low, mod, mod-high, high, very high risk) and PT failures (with, without PT failure); Relationship between 2 variables (FRS - each risk category, PT failure - with/without PT failure) expressed as a p-value
Statistical Analysis 2: Comparison: CAC Risk Category; CAC risk categories (low, low-moderate, mod -high, high, and very high); Test type: Other; p = 0.49, Fisher Exact — Relationship between CAC and PT failures. CAC risk category (low, low-mod, mod-high, high, very high risk) and PT failures (with, without PT failure); Relationship between 2 variables (CAC - each risk category, PT failure - with/without PT failure) expressed as a p-value

7. Secondary Outcome: Years of Military Service - Compare FRS to CAC
Description: Compare FRS category to CAC risk category for those with 10-14, 15-19, 20-24 and 25+ years of military service. Calculate Fisher's Exact test statistic and associated p values to look at the relationship between those with 10-14, 15-19, 20-24 and 25+ years of military service and FRS & CAC risk category. The CAC risk category (scale) = CAC score (estimated degree of calcium in coronary arteries, a number) + percentage by age to establish risks of future CV events. There are 5 risk categories: low, low - moderate, moderate - high, very high. The Framingham risk category (scale) = FRS to estimate the risk of a CV event over the next 10 years. The FRS uses age, systolic blood pressure, high-density lipoprotein and total cholesterol levels, and smoking status to create a score that is converted into a 10-year CV disease risk % that correlates into a risk category: low, moderate, moderate - high risk, very high. For both scales, low is the best and very high is the worst outcome
Time Frame: within 10 days of CT scan
Population: Unable to perform statistical test for 10-14 years of service due to small number of subjects (7). Data are separated into 4 rows (groups). Participants were placed into 1 of 4 groups based on certain criteria. Each group has a different number of participants. The total for all groups (rows) is equal to the overall number of participants analyzed
Measure: Count of Participants; unit: Participants
Groups:
- FRS Risk Category: Compare FRS risk categories (low, moderate, moderate -high, high, and very high) among groups
- CAC Risk Category: Compare CAC risk categories (low, low - moderate, moderate -high, high, and very high) among groups
Arm/Group | FRS Risk Category | CAC Risk Category
Number analyzed (Participants) | 100 | 100
Participants
  15-19 years of military service: number analyzed (Participants) | 44 | 44
  15-19 years of military service: low risk | 40 | 0
  15-19 years of military service: low - moderate / moderate risk | 0 | 40
  15-19 years of military service: moderate - high | 4 | 1
  15-19 years of military service: high risk | 0 | 3
  15-19 years of military service: very high risk | 0 | 0
  20-24 years of military service: number analyzed (Participants) | 40 | 40
  20-24 years of military service: low risk | 39 | 0
  20-24 years of military service: low - moderate / moderate risk | 1 | 35
  20-24 years of military service: moderate - high | 0 | 1
  20-24 years of military service: high risk | 0 | 3
  20-24 years of military service: very high risk | 0 | 1
  25 or more years of military service: number analyzed (Participants) | 16 | 16
  25 or more years of military service: low risk | 14 | 0
  25 or more years of military service: low - moderate / moderate risk | 0 | 9
  25 or more years of military service: moderate - high | 2 | 6
  25 or more years of military service: high risk | 0 | 0
  25 or more years of military service: very high risk | 0 | 1
Statistical Analysis 1: Comparison: FRS Risk Category; FRS risk categories (low, moderate, moderate -high, high, and very high); Test type: Other; p = 0.11, Fisher Exact — Relationship between FRS and overall years of service. FRS risk category (low, mod, mod-high, high, very high risk) and overall years of service (15-19, 20-24, 25+); Relationship between 2 variables (FRS - each risk category, overall years of service) expressed as a p-value
Statistical Analysis 2: Comparison: CAC Risk Category; CAC risk category (low, low-mod, mod-high, high, very high risk); Test type: Other; p = 0.003, Fisher Exact — Relationship between CAC and overall years of service. CAC risk category (low, low-mod, mod-high, high, very high risk) and overall years of service (15-19, 20-24, 25+); Relationship between 2 variables (CAC - each risk category, overall years of service) expressed as a p-value

8. Secondary Outcome: Additional Cardiovascular Risk Factors - Compare FRS to CAC
Description: Compare FRS category to CAC risk category for those with 1 risk factor (RF), vs 2 RF, vs 3 RF, vs 4 RF, vs 5 CV risk factors. Calculate Fisher's Exact test statistic and associated p values to look at the relationship between those with 1 RF, vs 2 RF, vs 3 RF, vs 4 RF, vs 5 CV RF and the FRS & CAC risk category. The CAC risk category (scale) = CAC score (estimated degree of calcium in coronary arteries, a number) + percentage by age to establish risks of future CV events. There are 5 risk categories: low, low - moderate, moderate - high, very high. The Framingham risk category (scale) = FRS to estimate the risk of a CV event over the next 10 years. The FRS uses age, systolic blood pressure, high-density lipoprotein and total cholesterol levels, and smoking status to create a score that is converted into a 10-year CV disease risk % that correlates into a risk category: low, moderate, moderate - high risk, very high. For both scales, low is the best and very high is the worst outcome
Time Frame: within 10 days of CT scan
Population: No data collected for this analysis. Due to the relatively small sample size with positive CAC scores, sub-analyses for patients with 2 or more risk factors were not performed. This may be an area for investigation if a larger study population were enrolled
Arm/Group | FRS Risk Category | CAC Risk Category
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Metabolic Syndrome - CAC
Description: Compare CAC risk category between two groups, those that meet criteria for metabolic syndrome and those that do not, to see if there is an association between the groups and CAC risk category. The number of participants in each risk category will be added. Then the total number for each group will be used to calculate the correlation using Fisher's Exact test and reported as a p value. The CAC risk category (scale) = CAC score (estimated degree of calcium in coronary arteries, a number) + percentage by age to establish risks of future CV events. There are 5 risk categories: low, low - moderate, moderate - high, high, very high. Low risk is the best outcome, and very high risk is the worst
Time Frame: within 10 days of CT scan
Population: The data is separated into two rows. Each row corresponds to a group. Participants were placed into one of the two groups based on certain criteria. Each group has a different number of participants analyzed. The total for both groups (rows) is equal to the overall number of participants analyzed
Measure: Count of Participants; unit: Participants
Groups:
- Coronary Artery Calcification (CAC): Compare CAC risk categories (low, low-mod, mod-high, high and very high) between groups
Arm/Group | Coronary Artery Calcification (CAC)
Number analyzed (Participants) | 107
Participants
  metabolic syndrome: number analyzed (Participants) | 23
  metabolic syndrome: low risk | 0
  metabolic syndrome: low - moderate risk | 18
  metabolic syndrome: moderate - high risk | 4
  metabolic syndrome: high risk | 1
  metabolic syndrome: very high risk | 0
  no metabolic syndrome: number analyzed (Participants) | 84
  no metabolic syndrome: low risk | 0
  no metabolic syndrome: low - moderate risk | 73
  no metabolic syndrome: moderate - high risk | 4
  no metabolic syndrome: high risk | 5
  no metabolic syndrome: very high risk | 2
Statistical Analysis 1: Comparison: Coronary Artery Calcification (CAC); CAC risk category (low, low-mod, mod-high, high, very high); Test type: Other; p = 0.21, Fisher Exact — [p-value comment as in outcome 4, analysis 2]; [statistical method as in outcome 4, analysis 2]

10. Secondary Outcome: Living in the Doors - CAC
Description: Compare CAC risk category between two groups, those who lived in the dorm for > 5 years and < 5 years, to see if there is an association between the groups and CAC risk category. The number of participants in each risk category will be added. Then the total number for each group will be used to calculate the correlation using Fisher's Exact test and reported as a p value. The CAC risk category (scale) = CAC score (estimated degree of calcium in coronary arteries, a number) + percentage by age to establish risks of future CV events. There are 5 risk categories: low, low - moderate, moderate - high, high, very high. Low risk is the best outcome, and very high risk is the worst outcome
Time Frame: within 10 days of CT scan
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary Artery Calcification (CAC)
Number analyzed (Participants) | 107
Participants
  > 5 years living in dorms: number analyzed (Participants) | 10
  > 5 years living in dorms: low risk | 0
  > 5 years living in dorms: low - moderate risk | 7
  > 5 years living in dorms: moderate - high risk | 1
  > 5 years living in dorms: high risk | 2
  > 5 years living in dorms: very high risk | 0
  < 5 years living in dorms: number analyzed (Participants) | 97
  < 5 years living in dorms: low risk | 0
  < 5 years living in dorms: low - moderate risk | 84
  < 5 years living in dorms: moderate - high risk | 7
  < 5 years living in dorms: high risk | 4
  < 5 years living in dorms: very high risk | 2
Statistical Analysis 1: Comparison: Coronary Artery Calcification (CAC); CAC risk category (low, low-mod, moderate - high, high, and very high); Test type: Other; p = 0.13, Fisher Exact — [p-value comment as in outcome 5, analysis 2]; [statistical method as in outcome 5, analysis 2]

11. Secondary Outcome: PT Failures - CAC
Description: Compare CAC risk category between two groups, those with and without a PT failures, to see if there is an association between the groups and CAC risk category. The number of participants in each risk category will be added. Then the total number for each group will be used to calculate the correlation using Fisher's Exact test and reported as a p value. The CAC risk category (scale) = CAC score (estimated degree of calcium in coronary arteries, a number) + percentage by age to establish risks of future CV events. There are 5 risk categories: low, low - moderate, moderate - high, very high. Low risk is the best outcome, and very high risk is the worst outcome
Time Frame: within 10 days of CT scan
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Coronary Artery Calcification (CAC)
Number analyzed (Participants) | 106
Participants
  with PT failures: number analyzed (Participants) | 53
  with PT failures: low risk | 0
  with PT failures: low - moderate risk | 46
  with PT failures: moderate - high risk | 3
  with PT failures: high risk | 2
  with PT failures: very high risk | 2
  without PT failures: number analyzed (Participants) | 53
  without PT failures: low risk | 0
  without PT failures: low - moderate risk | 44
  without PT failures: moderate - high risk | 5
  without PT failures: high risk | 4
  without PT failures: very high risk | 0
Statistical Analysis 1: Comparison: Coronary Artery Calcification (CAC); CAC risk categories (low, low-moderate, mod -high, high, and very high); Test type: Other; p = 0.49, Fisher Exact — [p-value comment as in outcome 6, analysis 2]; [statistical method as in outcome 6, analysis 2]

12. Secondary Outcome: Years of Military Service - CAC
Description: Compare CAC risk category among groups, those with 10-14, 15-19, 20-24, and 25+ years of military service, to see if there is an association between overall years of military service and CAC risk category. The number of participants in each risk category will be added. Then the total number for each group will be used to calculate the correlation using Fisher's Exact test and reported as a p value. The CAC risk category (scale) = CAC score (estimated degree of calcium in coronary arteries, a number) + percentage by age to establish risks of future CV events. There are 5 risk categories: low, low - moderate, moderate - high, very high. Low risk is the best outcome, and very high risk is the worst outcome
Time Frame: within 10 days of CT scan
Population: The data is separated into 4 rows. Each row corresponds to a group. Participants were placed into one of the 4 groups based on certain criteria. Each group has a different number of participants analyzed. The total for all groups (rows) is equal to the overall number of participants analyzed
Measure: Count of Participants; unit: Participants
Groups:
- Coronary Artery Calcification (CAC): Compare CAC risk categories (low, low-mod, mod-high, high and very high) among groups
Arm/Group | Coronary Artery Calcification (CAC)
Number analyzed (Participants) | 107
Participants
  10-14 years of military service: number analyzed (Participants) | 7
  10-14 years of military service: low risk | 0
  10-14 years of military service: low - moderate risk | 7
  10-14 years of military service: moderate - high risk | 0
  10-14 years of military service: high risk | 0
  10-14 years of military service: very high risk | 0
  15-19 years of military service: number analyzed (Participants) | 44
  15-19 years of military service: low risk | 0
  15-19 years of military service: low - moderate risk | 40
  15-19 years of military service: moderate - high risk | 1
  15-19 years of military service: high risk | 3
  15-19 years of military service: very high risk | 0
  20-24 years of military service: number analyzed (Participants) | 40
  20-24 years of military service: low risk | 0
  20-24 years of military service: low - moderate risk | 35
  20-24 years of military service: moderate - high risk | 1
  20-24 years of military service: high risk | 3
  20-24 years of military service: very high risk | 1
  25 or more years of military service: number analyzed (Participants) | 16
  25 or more years of military service: low risk | 0
  25 or more years of military service: low - moderate risk | 9
  25 or more years of military service: moderate - high risk | 6
  25 or more years of military service: high risk | 0
  25 or more years of military service: very high risk | 1
Statistical Analysis 1: Comparison: Coronary Artery Calcification (CAC); CAC risk category (low, low-mod, mod-high, high, very high risk); Test type: Other; p = 0.003, Fisher Exact — [p-value comment as in outcome 7, analysis 2]; Relationship between 2 variables (CAC - each risk category, overall years of service) expressed as a p-value

13. Secondary Outcome: Additional Risk Factors - CAC
Description: Compare CAC risk category among groups, those with 1 risk factor (RF) vs. 2 RF, vs 3 RF, vs 4 RF, vs 5 RF (as listed in the inclusion criteria), to see if there is an association between the groups and CAC risk category. The number of participants in each risk category will be added. Then the total number for each group will be used to calculate the correlation using Fisher's Exact test and reported as a p value. The CAC risk category (scale) = CAC score (estimated degree of calcium in coronary arteries, a number) + percentage by age to establish risks of future CV events. There are 5 risk categories: low, low - moderate, moderate - high, very high. Low risk is the best outcome, and very high risk is the worst outcome
Time Frame: within 10 days of CT scan
Population: as for outcome 8
Arm/Group | Coronary Artery Calcification (CAC)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: through study completion, up to 10 days
Groups:
- Compare CAC and FRS: Coronary Artery Calcium (CAC) scores are reported as a numerical value and a percentage for age that is then regarded in terms of risk categories. The Framingham Risk Score (FRS) is a standard of care for estimating risk of a cardiovascular event over the next 10 years
Arm/Group | Compare CAC and FRS
All-Cause Mortality (participants affected / at risk) | 0/104
Serious Adverse Events (participants affected / at risk) | 0/104
Other Adverse Events (participants affected / at risk) | 0/104

LIMITATIONS AND CAVEATS:
There were only 3 female participants; therefore, generalizations could not be made for this gender

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/30/NCT02009930/Prot_SAP_000.pdf